CLINICAL TRIAL: NCT00361192
Title: Sensitivity and Specificity of Color Doppler Directed Temporal Artery Biopsy as Compared to Standard Random Biopsy in the Diagnosis of Temporal Arteritis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TEMP ARTERITIS 001A
Record Dates: First submitted 2006-08-06; First posted 2006-08-08 (Estimated); Last update posted 2006-12-06 (Estimated); Status verified 2006-08

CONDITIONS: Temporal Arteritis; Duplex of Temporal Artery; Biopsy of Temporal Artery
Keywords: temporal arteritis; duplex of temporal artery; biopsy of temporal artery
MeSH Terms: conditions — Giant Cell Arteritis

INTERVENTIONS:
Procedure: biopsy of temporal artery

SUMMARY:
Introduction

Temporal arteritis (TA) is the most common primary vasculitis in the adult population. TA is a systemic multi-organ disease but primarily involves the cranial arteries, especially the temporal artery. The signs and symptoms of the disease are variable and therefore the differential diagnosis is often difficult. The annual incidence of the disease in the population above the age of 50 in Jerusalem is about 10 per 100,000.

Diagnosis is based on the clinical findings and confirmed by biopsy of the temporal artery, positive for histologic findings of arteritis. Though the biopsy procedure is minor and can be accomplished under local anesthesia, it is not without morbidity. Along with minor pain, more serious complications - facial nerve injury, ptosis, stroke, and local necrosis of skin - have been reported.

A negative biopsy does not completely rule out the diagnosis of TA because of the segmental nature of the inflammation. Even if one removes an appropriate length of artery (usually 1-2 cm) the possibility exists that an involved segment may not have been included and the biopsy will be reported as normal.

It has recently been reported that color Doppler ultrasonography can be used to diagnose TA. Arterial inflammation causing peri-vascular edema appearing as a "dark halo" and segmental stenosis of the temporal artery are characteristic ultrasound findings suggestive of TA. If there is no dark halo sign, a diagnosis of TA cannot be supported and temporal artery biopsy can be avoided in most of these patients. The presence of the dark halo sign has a positive predictive value of only 50%.

As noted above the disease is characterized by segmental involvement of the artery and to avoid a false negative biopsy, excision of up to 3cm of the artery has been recommended, thereby increasing the morbidity, and leading patients to refuse the procedure. Use of ultrasound-guided biopsy of the artery may dramatically raise the sensitivity and specificity of the biopsy and reduce the requirement for excising long segments of artery.

Objective

The objective of this study is to examine the use of ultrasound-guided biopsy of the temporal artery in the diagnosis of TA. Ultrasound-guided biopsy will be compared to the standard random biopsy generally in use. Appropriate statistical methods will be employed.

Methods

The Vascular Laboratory in Shaare Zedek Medical Center performs approximately 200 Doppler ultrasound studies of the temporal artery each year at the request of community-based physicians. Some of these patients are then also referred for biopsy of the temporal artery at various surgical facilities in the city. In collaboration with the referring physician, the patients will be offered a combined diagnostic Doppler ultrasound and guided biopsy on the basis of clinical guidelines and according to the ultrasound findings as described below.

Patients suffering from signs and symptoms consistent with TA and who have not undergone previous temporal artery biopsy will be included.

Patients suffering from isolated polymyalgia rheumatica will be excluded. Patients who are already undergoing steroid treatment will be excluded. Patients with an ultrasound study that is positive for the dark halo sign will be divided into two groups on a random basis after obtaining informed consent.

One group will undergo ultrasound-guided biopsy, while the other will undergo biopsy as is the standard practice in our institution - a 1-2cm length of temporal artery will be excised from the preauricular area.

If the ultrasound is negative, no biopsy will be done in the setting of this study.

It is expected that about 50 patients will be accrued during the 6-month study period. Differences in outcome will be analyzed using Fishers exact test.

Approval from the Helsinki committee of Shaare Zedek Medical Center has been requested.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from signs and symptoms consistent with TA and who have not undergone previous temporal artery biopsy will be included.

Exclusion Criteria:

* Patients suffering from isolated polymyalgia rheumatica will be excluded.
* Patients who are already undergoing steroid treatment will be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-08; Study Completion 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: David Shemesh, MD, Study Director — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel